CLINICAL TRIAL: NCT05746910
Title: Patient's Perception of Exercise After Bone Tumor Resection-A Qualitative Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Emel Mete, research assistant, Istanbul Medeniyet University
Other Study IDs: 2022/0179-1
Record Dates: First submitted 2023-02-17; First posted 2023-02-28 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Bone Cancer Tumor
Keywords: bone cancer tumor; exercise; Patient
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to investigate the opinions of patients who have undergone bone tumor resection surgery about post-op exercises.

DETAILED DESCRIPTION:
Semi-structured in-depth individual interviews will be conducted with patients who have undergone bone tumor surgery. In in-depth individual interviews, the same questions will be asked to all participants and the verbal answers to these questions will be recorded with voice recorders. Compared to taking notes by hand; It will be preferable to record the conversation with a voice recorder because it has advantages such as recording all the interviews and allowing the interviewer to focus on the interview. Thematic analysis method will be used in the evaluation of the data.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged between 18 and 65,
* Individuals without communication problems,
* Individuals who have been diagnosed with a bone tumor for the first time and who have undergone resection surgery
* Patients who have previously received therapeutic exercises

Exclusion Criteria:

* Uncontrollable arrhythmia and/or hypertension
* Presence of advanced sensory deficit
* Visual and hearing problems
* Not having sufficient communication skills (Mini-Mental Test score below 24 points)
* Patients undergoing head and neck bone resection

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Individuals who have been diagnosed with a bone tumor for the first time and who have undergone resection surgery
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2022-12-05 (Actual); Primary Completion 2023-03-30 (Estimated); Study Completion 2023-04-10 (Estimated)

PRIMARY OUTCOMES:
Semi-structured in-depth individual interviews about Patient's Perceptions of post-op exercises | baseline
  Semi-structured in-depth individual interviews will be conducted with patients only once. The same questions will be asked to all participants and the verbal answers to these questions will be recorded with voice recorders.

CONTACTS AND LOCATIONS:
Locations (1):
- Emel Mete, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No